CLINICAL TRIAL: NCT04599231
Title: Effects of Preoperative Anxiety and Depression on Short-term Postoperative Recovery Among Early Gastric Cancer Patients Undergoing Laparoscopic Gastrectomy
Brief Title: Effects of Preoperative Anxiety and Depression on Short-term Postoperative Recovery in Early Gastric Cancer
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Considering the various conditions (other ongoing prospective studies, lack of manpower), we decided not to proceed with this study.
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Hojin Lee, MD, Clinical assistant professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2008-130-1149
Record Dates: First submitted 2020-10-06; First posted 2020-10-22 (Actual); Last update posted 2022-12-07 (Actual); Status verified 2022-12

CONDITIONS: Postoperative Complications; Anxiety; Depression; Coping Behavior
Keywords: Postoperative Complications; Anxiety; Depression; Coping Behavior
MeSH Terms: conditions — Postoperative Complications; Anxiety Disorders; Depression

STUDY DESIGN:
Intervention Model Description: Prospective observational study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study group (Experimental): The investigators would perform the following tests preoperatively on the study subjects.
  1. Hospital Anxiety and Depression Scale (HADS)
  2. Amsterdam Preoperative Anxiety and Information Scale (APAIS)
  3. Coping and Adaptation Processing Scale-Short Form (CAPS-SF)
  4. Quality of Recovery -15 (QOR-15)
  Interventions: Diagnostic Test: Quality of Recovery -15

INTERVENTIONS:
Diagnostic Test: Quality of Recovery -15 — The investigators plan to evaluate patients' quality of recovery at postoperative day (POD) 1, 2, and 3.

SUMMARY:
This study aims to investigate preoperative anxiety, depression, and coping strategy of the patients undergoing laparoscopic gastrectomy for early gastric cancer and their effects on short-term postoperative recovery measured by Quality of Recovery-15 (QOR-15). The findings of the study would improve the perioperative management of early gastric cancer patients.

DETAILED DESCRIPTION:
The researchers plan to investigate preoperative psychological factors such as anxiety, depression, and coping strategy in association with short-term quality of recovery from surgery in 100 patients scheduled for early gastric cancer surgery (laparoscopic gastrectomy).

The following items are investigated before surgery; Age, sex, BMI, level of education, occupation, marital status, ECOG performance status, ASA physical status, Apfel score, history of mental disorder, type of surgery, past surgical history, the number of days from diagnosis of cancer to surgery, clinical stage of cancer, histological type of cancer, presence of chronic pain, Quality of Recovery-15 (QOR-15), Hospital Anxiety and Depression Scale (HADS), Amsterdam Preoperative Anxiety and Information Scale (APAIS), Coping and Adaptation Scale-Short Form (CAPS-SF).

The QOR-15 is investigated for 24, 48, and 72 hours after surgery. The severity of postoperative pain by the 11-point Numerical Rating Scale (NRS) is concurrently measured at 24, 48, and 72 hours after surgery. In addition, the researchers measure postoperative complications, particularly nausea/vomiting, at 24, 48, and 72 hours after surgery and length of stay by counting the number of days from the day of surgery to discharge.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or above
* Patients scheduled for early gastric cancer surgery (laparoscopic gastrectomy) under general anesthesia
* ASA status I or II
* Able to read and understand the information sheet, the questionnaires, and the consent form.

Exclusion Criteria:

* Unable to read and understand the information sheet, the questionnaires, and the consent form.
* Age above 80 years
* WIth severe medical or psychological diseases

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-10-12 (Estimated); Primary Completion 2021-06-24 (Estimated); Study Completion 2021-08-24 (Estimated)

PRIMARY OUTCOMES:
Quality of Recovery -15 score at postoperative 72 hours | at postoperative 72 hours
  There are total 15 items where each of them is an 11-point numerical rating scale (for positive items, 0 = "none of the time" to 10 = "all of the time"; for negative items, the scoring was reversed; maximum score 150)

SECONDARY OUTCOMES:
Quality of Recovery -15 score at postoperative 24 hours | at postoperative 24 hours
  There are total 15 items where each of them is an 11-point numerical rating scale (for positive items, 0 = "none of the time" to 10 = "all of the time"; for negative items, the scoring was reversed; maximum score 150)
Quality of Recovery -15 score at postoperative 48 hours | at postoperative 48 hours
  There are total 15 items where each of them is an 11-point numerical rating scale (for positive items, 0 = "none of the time" to 10 = "all of the time"; for negative items, the scoring was reversed; maximum score 150)
Postoperative pain score | at postoperative 24, 48, and 72 hours
  11-pointed NRS pain score at resting/coughing/movement NRS (0-10): 0, "no pain"; 10, "worst pain imaginable"
Length of stay | through study completion, an average of 1 year
  The number of days that patients spend in the hospital after surgery
Postoperative nausea or vomiting | at postoperative 24, 48, and 72 hours
  Patients' postoperative nausea/vomiting: for each, 0, no; 1 yes, but not severe enough to take antiemetics; 2, yes, severe enough to take antiemetics

CONTACTS AND LOCATIONS:
Overall Officials: Hojin Lee, MD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Background] Yoon S, Joo H, Oh YM, Lee J, Bahk JH, Lee HJ. Validation and clinical utility of the Korean version of the Quality of Recovery-15 with enhanced recovery after surgery: a prospective observational cohort study. Br J Anaesth. 2020 Oct;125(4):614-621. doi: 10.1016/j.bja.2020.06.040. Epub 2020 Jul 21. PMID 32703550
- [Background] Stark PA, Myles PS, Burke JA. Development and psychometric evaluation of a postoperative quality of recovery score: the QoR-15. Anesthesiology. 2013 Jun;118(6):1332-40. doi: 10.1097/ALN.0b013e318289b84b. PMID 23411725